CLINICAL TRIAL: NCT00074711
Title: Bone Sparing by Calcium Salts With and Without Extra Phosphorus
Brief Title: Adding Phosphorus to Osteoporosis Drug Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AR048846 (NIH); R01AR048846 (NIH)
Record Dates: First submitted 2003-12-19; First posted 2003-12-22 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Bone Mineral Density; Calcium
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Calcium Carbonate; calcium phosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium Phosphate Treatment Group (Active Comparator): Participants will receive teriparatide and vitamin D during the course of the 12-month study. They will also receive calcium phosphate.
  Interventions: Drug: Calcium Phosphate
- Calcium Carbonate Treatment Group (Active Comparator): Participants will receive teriparatide and vitamin D during the course of the 12-month study. They will also receive calcium carbonate.
  Interventions: Drug: Calcium carbonate

INTERVENTIONS:
Drug: Calcium carbonate — Participants will receive teriparatide and vitamin D during the course of the 12-month study. They will also receive calcium carbonate.
  Arms: Calcium Carbonate Treatment Group
Drug: Calcium Phosphate — Participants will receive teriparatide and vitamin D during the course of the 12-month study. They will also receive calcium phosphate.
  Arms: Calcium Phosphate Treatment Group

SUMMARY:
Osteoporosis causes bones to weaken and break more easily. Calcium and phosphorus are two minerals that are essential for normal bone formation. Unfortunately, calcium salts commonly prescribed in anti-osteoporosis treatment bind phosphorus from food and restrict phosphorus available for bone building. Teriparatide is a drug that reduces the risk of fractures by increasing bone thickness and strength. Vitamin D is also necessary for strong bones and teeth. The purpose of this study is to evaluate the bone-building effectiveness of two calcium supplements, one with a source of phosphorus and one without, in combination with teriparatide and vitamin D in women with osteoporosis.

DETAILED DESCRIPTION:
Osteoporosis is the most common type of bone disease. Calcium supplements normally used in anti-osteoporosis treatment are calcium salts of carbonate or citrate; however, these salts bind phosphorus from food in the intestine and restrict phosphorus available for bone building. This study will evaluate the efficacy of adding calcium phosphate to a regimen of teriparatide and vitamin D in increasing bone mineral density in women with osteoporosis. It is hypothesized that the group taking the phosphate-containing calcium supplement will have greater gains in bone mineral density (BMD) during the course of the study than the group not receiving phosphate.

All participants will receive teriparatide and vitamin D during the course of the 12-month study. Participants will be randomly assigned to one of two groups. One group will receive calcium phosphate and the other will receive calcium carbonate. BMD will be measured at spine and hip at baseline and at 3, 6, and 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Bone mineral density (BMD) T-score less than -1.0
* One or more vertebral fractures
* Serum creatinine less than 1.3 mg/dL
* Serum phosphorus less than 3.6 mg/dL
* Daily phosphorus intake below NHANES-III median
* Body mass index (BMI) less than 30 kg/m2

Exclusion Criteria:

* Paget's disease or history of osteosarcoma
* Systemic corticosteroid therapy
* Hyperparathyroidism
* Recent history of kidney stone
* Anticonvulsant therapy known to alter vitamin D metabolism
* Radiation therapy to bone

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2004-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Heaney, MD, Principal Investigator — Creighton University Medical Center
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Result] Heaney RP, Recker RR, Watson P, Lappe JM. Phosphate and carbonate salts of calcium support robust bone building in osteoporosis. Am J Clin Nutr. 2010 Jul;92(1):101-5. doi: 10.3945/ajcn.2009.29085. Epub 2010 May 19. PMID 20484446
- [Derived] Heaney RP, Watson P. Variability in the measured response of bone to teriparatide. Osteoporos Int. 2011 Jun;22(6):1703-8. doi: 10.1007/s00198-010-1376-1. Epub 2010 Sep 9. PMID 20827548

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcium Phosphate Treatment Group | Calcium Carbonate Treatment Group
Started | 120 | 121
Completed | 105 | 106
Not Completed | 15 | 15
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 10 | 8
Not completed — Participant stopped study drug | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium Phosphate Treatment Group | Calcium Carbonate Treatment Group | Total
Number analyzed (Participants) | 120 | 121 | 241
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 115 | 115 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.09 (7.02) | 70.07 (6.34) | 70.07 (6.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 121 | 241
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 120 | 121 | 241

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Spine and Hip BMD, Measured as Grams Per Square Centimeter.
Description: Bone mineral density (BMD, measured by dual X-ray absorptiometry - DEXA) measured at several intervals during the study. BMD measured as grams per square centimeter (g/cm2).
Time Frame: Measured at Baseline
Population: Postmenopausal women with spinal osteoporosis.
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Calcium Phosphate Treatment Group | Calcium Carbonate Treatment Group
Number analyzed (Participants) | 105 | 106
g/cm2
  Baseline (Hip) | 0.76 (0.11) | 0.78 (0.10)
  Baseline (Spine) | 0.88 (0.12) | 0.86 (0.12)

2. Primary Outcome: Bone Mineral Density (BMD) Under Treatment With an Anabolic Agent (Teriparatide).
Description: The principle outcome measure was change in bone mineral density (BMD) under treatment with an anabolic agent (teriparatide).
Time Frame: 12 months
Population: Participants that completed study.
Measure: Mean (Standard Error); unit: g/cm2
Arm/Group | Calcium Phosphate Treatment Group | Calcium Carbonate Treatment Group
Number analyzed (Participants) | 105 | 106
g/cm2
  Hip Bone Mineral Density | 0.01680 (0.00227) | 0.01450 (0.00203)
  Spine Bone Mineral Density | 0.0609 (0.00356) | 0.0607 (0.00336)

3. Secondary Outcome: Change From Baseline in Serum Phosphorus, Serum Creatinine, Serum Calcium at 12 Months
Time Frame: Measured at baseline and 12 months
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Calcium Phosphate Treatment Group | Calcium Carbonate Treatment Group
Number analyzed (Participants) | 105 | 106
mg/dl
  S Phos | 0.139 (0.045) | 0.245 (0.042)
  S Crt | -0.001 (0.012) | 0.051 (0.012)
  S Ca | -0.048 (0.041) | 0.001 (0.047)

4. Secondary Outcome: Change From Baseline in Urinary Calcium to Creatinine Ratio, Urinary Phosphorus to Creatinine Ratio at 12 Months
Time Frame: Measured at baseline and 12 months
Measure: Mean (Standard Error); unit: g/g
Arm/Group | Calcium Phosphate Treatment Group | Calcium Carbonate Treatment Group
Number analyzed (Participants) | 105 | 106
g/g
  Ca to CRT | 0.021 (0.010) | 0.011 (0.010)
  Ph to CRT | 0.073 (0.025) | -0.053 (0.028)

5. Secondary Outcome: Change From Baseline in Urinary N-telopeptide at 12 Months
Time Frame: Measured at baseline and 12 months
Measure: Mean (Standard Error); unit: nmol bce/mmol
Arm/Group | Calcium Phosphate Treatment Group | Calcium Carbonate Treatment Group
Number analyzed (Participants) | 105 | 106
nmol bce/mmol | 16.0 (3.42) | 17.1 (2.79)

6. Secondary Outcome: Change From Baseline in Urinary Hydroxyproline to Creatinine Ratio at 12 Months
Time Frame: Measured at baseline and 12 months
Measure: Mean (Standard Error); unit: micromol/mmol
Arm/Group | Calcium Phosphate Treatment Group | Calcium Carbonate Treatment Group
Number analyzed (Participants) | 105 | 106
micromol/mmol | 5.61 (1.25) | 6.26 (0.962)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Calcium Phosphate Treatment Group | Calcium Carbonate Treatment Group
Serious Adverse Events (participants affected / at risk) | 1/105 | 0/106
Other Adverse Events (participants affected / at risk) | 0/105 | 0/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcium Phosphate Treatment Group (N=105) | Calcium Carbonate Treatment Group (N=106)
Death (Cardiac disorders) | 1 (1) | 0 (0) — Death was judged by the DSMB to be unrelated to the study or its components

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No